CLINICAL TRIAL: NCT00500695
Title: Enhancing Motivation To Quit Smoking In Smokers With Serious Mental Illness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marc L. Steinberg, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 220045018; K23DA018203 (NIH)
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing (Experimental): Motivational Interviewing
  Interventions: Behavioral: Motivational Interviewing
- Psychoeducation (Active Comparator): Psychoeducation
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational Interviewing
  Arms: Motivational Interviewing
Behavioral: Psychoeducation — Psychoeducation
  Arms: Psychoeducation

SUMMARY:
This project will assess the utility of a brief motivational intervention to engage smokers with schizophrenia in treatment for tobacco dependence treatment. It is hypothesized that a brief motivational intervention will be more effective in engaging smokers with schizophrenia to tobacco dependence treatment than an educational intervention. The educational intervention will increase the likelihood to reducing cigarette intake and/or attending tobacco dependence treatment by teaching subjects about the negative effects of smoking and the success of tobacco dependence treatment. The motivational intervention will increase the likelihood to reducing cigarette intake and/or attending tobacco dependence treatment by increasing subjects' motivation to change by presenting objective and personalized information regarding their smoking behaviors in a non-judgmental and supportive manner.

DETAILED DESCRIPTION:
See Brief Summary above.

ELIGIBILITY:
Inclusion Criteria:

* Current smokers must be over the age of 18,
* Must have a diagnosis of schizophrenia or schizoaffective disorder
* Must smoke at least 10 cigarettes per day
* Must be capable of giving informed consent as measured by Folstein Mini Mental Status Exam of at least 22

Exclusion Criteria:

•Those unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Attendance at first smoking cessation session | one month

SECONDARY OUTCOMES:
Cigarettes per day | 1-Month Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: Marc L. Steinberg, PH.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ- Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States